CLINICAL TRIAL: NCT07248631
Title: Combined Effects of Foot-Ankle Therapeutic Exercises and Mindful Walking on Pain, Foot and Ankle Disability and Quality of Life in Patients With Diabetic Polyneuropathy
Brief Title: Combined Effects of Foot-Ankle Therapeutic Exercises and Mindful Walking in Patients With Diabetic Polyneuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/02104 Ayesha Ahsan Kamal
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Polyneuropathy
Keywords: Pain; Quality of life; Foot-Ankle therapeutic Exercises; Mindful Walking; Diabetic Polyneuropathy; Foot and Ankle Disability
MeSH Terms: conditions — Diabetic Neuropathies; Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot-Ankle therapeutic exercises and Mindful Walking (Active Comparator): Participants will receive 12 weeks program of foot-ankle therapeutic exercises combined with mindful walking. The intervention arm will consist of an 12-weeks program combining foot-ankle therapeutic exercises and mindful walking. Participants will attend sessions three times a week, with each session lasting 30 minutes for both exercises and mindful walking. The foot-ankle therapeutic exercises will include strengthening exercises like toe spreads, toe curls, heel raises, and calf raises, as well as flexibility exercises such as ankle dorsiflexion stretch, plantar fascia stretch, and calf stretch. The exercises will progress in intensity and difficulty over the 12-week period. Mindful walking sessions will incorporate sensory cues, including kinesthetic, visual, auditory, and tactile cues. Assessments will be conducted at baseline and 12 weeks to evaluate pain, foot and ankle disability, and quality of life.
  Interventions: Other: Standard care with Mindful walking.
- Standard Care and Mindful Walking (Active Comparator): Participants will receive 12 weeks program of standard care combined with Mindful walking. Group 2 will receive standard care combined with mindful walking for 12 weeks. Participants will attend sessions three times a week, with each session lasting 30 minutes. The mindful walking sessions will incorporate sensory cues, including kinesthetic cues, visual cues, auditory cues, and tactile cues. The standard care will be provided alongside the mindful walking intervention. Assessments will be conducted at baseline and 8 weeks to evaluate pain, foot and ankle disability, and quality of life.
  Interventions: Other: Foot-Ankle therapeutic exercises and Mindful Walking.

INTERVENTIONS:
Other: Foot-Ankle therapeutic exercises and Mindful Walking. — The intervention consists of Foot-Ankle Therapeutic Exercises combined with Mindful Walking, specifically designed to address diabetic neuropathy symptoms. This 12-week program includes strengthening exercises such as toe spreads, toe curls, heel raises, calf raises, single leg stance, and ankle dorsiflexion, as well as flexibility exercises like ankle dorsiflexion stretch, plantar fascia stretch, calf stretch, toe flexion stretch, and Achilles tendon stretch. Alongside these exercises, participants will engage in mindful walking practices incorporating sensory cues (kinesthetic, visual, auditory, and tactile cues). The unique combination and structured progression of these exercises and mindfulness techniques distinguish this intervention from other therapeutic approaches.
  Arms: Standard Care and Mindful Walking
Other: Standard care with Mindful walking. — The intervention consists of Foot-Ankle Therapeutic Exercises combined with Mindful Walking, specifically designed to address diabetic neuropathy symptoms. This 12-week program includes strengthening exercises such as toe spreads, toe curls, heel raises, calf raises, single leg stance, and ankle dorsiflexion, as well as flexibility exercises like ankle dorsiflexion stretch, plantar fascia stretch, calf stretch, toe flexion stretch, and Achilles tendon stretch. Alongside these exercises, participants will engage in mindful walking practices incorporating sensory cues (kinesthetic, visual, auditory, and tactile cues). The unique combination and structured progression of these exercises and mindfulness techniques distinguish this intervention from other therapeutic approaches.
  Arms: Foot-Ankle therapeutic exercises and Mindful Walking

SUMMARY:
The aim of this study is to investigate the combined effects of foot ankle therapeutic exercises and mindful walking on pain, foot and ankle disability, and quality of life in patients with diabetic polyneuropathy. This study seeks to evaluate the efficacy of these interventions in improving clinical outcomes and enhancing the overall well-being of individuals with diabetic polyneuropathy.

DETAILED DESCRIPTION:
A 12-week foot-ankle therapeutic exercise program has been found to show positive effects compared to usual care on fast-gait speed, foot-ankle range of motion, vibration sensitivity, and quality of life in people with diabetic neuropathy.

Mindful walking's efficacy for chronic low back pain management has been investigated, with a randomized controlled trial of 55 patients yielding no significant improvements in pain intensity, back function, or stress after 8 weeks.

Exercise therapy has been found to significantly improve gait function in patients with diabetic peripheral neuropathy. A systematic review of 9 randomized controlled trials (370 participants) showed that exercise therapy enhances 6-minute walk test, 10-meter walk test, and Tinetti scale outcomes, improving mobility and reducing fall risk.

Exercise shows therapeutic potential for sensory nerve disorders, improving symptoms in most cases. Benefits are seen in diabetic pain and nerve damage, with varying mechanisms underlying these effects. Exercise therapy enhances outcomes for various nerve-related disorders, improving symptoms by at least two times compared to no exercise.

A 12-week study found significant improvements in glycemic control and vascular function in patients with type 2 diabetes who practiced Buddhist walking meditation, whereas traditional walking only improved blood glucose levels and cardiovascular fitness.

A study on sensor-based interactive balance training with visual joint movement feedback found significant improvements in postural stability in patients with diabetic peripheral neuropathy. The intervention group demonstrated a 62.68% reduction in CoM sway with eyes closed.

Physical therapy has been shown to impact limited joint mobility in diabetic neuropathy patients. A study found significant joint mobility improvements after 10 sessions of passive joint mobilization, with near-normal mobility achieved after 20 sessions.

A 4-week multimodal treatment program (treadmill, muscle strengthening, balance training) significantly improved gait endurance and functional independence in diabetic neuropathy patients, with sustained benefits at 2-month follow-up.

Foot biomechanics in diabetes mellitus patients has been studied, with an observational study of 281 patients finding no significant differences in joint mobility between patients with and without neuropathy.

Diabetic neuropathy significantly impairs ankle strength and balance recovery in older women, despite normal clinical muscle testing.

Despite the established benefits of exercise and physical therapy in managing diabetic polyneuropathy (DPN), significant knowledge gaps persist. Existing studies have primarily focused on isolated interventions, such as foot-ankle exercises or mindful walking, without exploring their combined effects. The synergistic potential of integrating therapeutic exercises with mindfulness-based walking remains uninvestigated. Insufficient evidence supports optimal exercise protocols and mindfulness-based interventions for DPN management. This study addresses these gaps, paving the way for evidence-based DPN management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetic polyneuropathy (DPN) confirmed by medical history and clinical examination.
* Experience pain and disability in foot/ankle, with a Numeric Pain Rating Scale (NPRS) score ≥ 4.
* Independent walking ability for at least 10 m.
* Age (40-75) years.
* Ability to understand and follow exercise instructions.
* A maximum of one amputated toe, not being the hallux.
* Willingness to participate in the study and provide informed consent.

Exclusion Criteria:

* Presence of an active plantar ulcer or gangrene.
* History of surgical procedure at the knee, ankle, or hip or indication of surgery throughout the intervention period.
* Arthroplasty and/or orthosis of lower limbs or indication of lower limb arthroplasty throughout the intervention period.
* Participating in other exercise programs or studies.
* Dementia or inability to give consistent information.
* Diagnosis of neurological diseases.
* Neuropathic pain due to other causes (e.g., HIV, chemotherapy).
* Major vascular complications and/or severe retinopathy.

Ages: 40 Months to 75 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | At baseline and 12 weeks
  The Numeric Pain Rating Scale (NRS) is scored by having a patient select a number from \(0\) to \(10\) to represent their pain level. A score of \(0\) indicates "no pain," while a score of \(10\) represents "the worst pain imaginable". The higher the number, the greater the intensity of the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Tariq, MS, Principal Investigator — Riphah International University
Locations (1):
- Nishtar 2, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No